CLINICAL TRIAL: NCT01758770
Title: Multi Center Survey on Spine and Hip Status in Chinese Population Using Quantitative Computed Tomography (QCT)
Brief Title: China Action on Spine and Hip Status
Acronym: CASH
Status: Completed | Type: Observational
Sponsor: Beijing Jishuitan Hospital (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other); University of California, San Francisco (Other); Beijing Shi Jing Shan hospital,Beijing, China (Unknown); Tai yuan central hospital,taiyuan, shanxi (Unknown); Cheng Du Da Yi hospital,Cheng du, Sichuan (Unknown); Shen Yang 4th hospital,shen yang, liaoning (Unknown); Second hospital of sichuan university,Cheng du, Sichuan (Unknown); Chang Zhou Wu Jin Traditional Chinese Medicine hospital (Unknown); Red cross hospital of Shaanxi (Unknown); No 1 TCM hospital of Jiangsu (Unknown); No 2 TCM hospital of Jiangsu (Unknown); Chengdu Second people's hospital (Unknown); Affiliate hospital of jiangxi Traditional Chinese Medicine university (Unknown)
Responsible Party: Principal Investigator, xiaoguang Cheng, Chairman, department of radiology, Beijing Jishuitan Hospital
Other Study IDs: jst2012cash
Record Dates: First submitted 2012-12-26; First posted 2013-01-01 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Osteoporosis; Liver Steatosis; Metabolic Syndrome; Obesity
Keywords: osteoporosis; osteoarthritis; bone mineral density; computed xray tomography; liver steatosis; obesity
MeSH Terms: conditions — Osteoporosis; Fatty Liver; Metabolic Syndrome; Obesity; Osteoarthritis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To determine the prevalences of osteoporotic fracture in elderly Chinese population.
2. To determine the prevalences of osteoporosis in elderly Chinese population using QCT BMD measurement.
3. To investigate the difference in the prevalences of osteoporosis between cities and urban-rural area in China.
4. To investigate the association of body composition with osteoporosis
5. To investigate the prevalence of liver steatosis in China
6. To investigate the application of QCT fat measurement

DETAILED DESCRIPTION:
Osteoporosis and osteoarthritis (OA) both are very common in elderly population,it is particular important for China with a huge aging population in the coming years.Bone mineral density measured by quantitative computed tomography (QCT) or dual energy X-ray absorptiometry (DXA) is the surrogate for bone health status and diagnosis of osteoporosis and OA. In this study we utilize the large-scale population based epidemiology study (PURE) population,spine and hip QCT and/or DXA will be obtained for the subject to investigate the prevalence of osteoporosis and osteoarthritis in elderly Chinese population. We also study the relation between bone mineral density with osteoporotic fracture and OA More than 3000 subjects selected from the PURE study participants in Beijing and other centers in China will be recruited to this study. More precisely, the subjects are consisted of the females over 55 years and males over 60 years old, along with the 20% randomly selected PURE participants for blood sampling.

Beijing ji shui tan hospital will be the coordinate center for the whole study, Beijing shi jing shan hospital, Beijing shun yi traditional medicine hospital and Taiyuan central hospital of shanxi will participate, other centers may be added late.

Bone mineral density of spine and hip will be measured with QCT and/or DXA. Quantitative computed tomography QCT pro (Mindways software, inc. USA) will be used for all QCT measurement, the CT scanner will be the clinical CT scanner of the local participated center.

Quality control and monitoring will be conducted by Beijing ji shui tan hospital, as well as the centralised image interpretation.

Therefore, this study is designed to provide the current and reliable prevalence of osteoporotic fracture, osteoporosis, OA in elderly Chinese population using QCT and/or DXA. The performance of QCT and DXA in the diagnosis of osteoporosis , as well as the association of body composition with osteoporosis will be assessed.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Participants of the PURE study in China (PURE China study)
   2. be willing to and be able to join in the study and signed Informed consent
2. Exclusion Criteria:

   1. Pregnant
   2. Spine and both hip implants

Ages: 29 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a population-based study, the population of this study is the subset of participants of the large-scale population-based study:the prospective urban rural epidemiology (PURE) in China.
Sampling Method: Non-Probability Sample
Enrollment: 3457 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Osteoporotic fractures | 5 years
  The spine osteoporotic fractures assessed on the lateral spine image of QCT exam
Bone mineral density (BMD) of spine and hip | 5 years
  BMD measurement at the spine by QCT and hip
liver steatosis | 5 years
  The liver steatosis assessed by QCT

SECONDARY OUTCOMES:
Metabolic syndrome | 5 years
  Diagnosis of metabolic syndrome and visceral fat
visceral fat measurement by QCT | 5 years
  visceral fat measurement and distribution assessed by QCT at the abdomen and hip
Osteoarthritis of spine and hip | 5 years
  OA assessment at spine and hip by CT images

CONTACTS AND LOCATIONS:
Overall Officials: xiaoguang cheng, MD, Principal Investigator — Beijing ji shui tan hospital
Locations (1):
- Beijing ji shui tan hospitla, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No